CLINICAL TRIAL: NCT05758610
Title: A Phase I Clinical Study of Safety, Tolerability, Pharmacokinetics, and Initial Efficacy of ETH-155008 Tablets in Patients With Relapsed or Refractory Acute Myeloid Leukemia and Non-Hodgkin's Lymphoma
Brief Title: A Phase I Study of Euthare-155008(ETH-155008) in AML and NHL Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shengke Pharmaceuticals (Jiangsu) Limited, China (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETH-155008- 101
Record Dates: First submitted 2023-02-15; First posted 2023-03-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: NHL, Adult; AML, Adult Recurrent
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Myeloid, Acute; Recurrence | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ETH-155008 (Experimental): Dose level: 20mg/day, 40mg/day, 60mg/day, 80mg/day, 100mg/day. Each dose level will recruit 1-6 subjects, taking ETH-155008 tablets once daily.
  Intervention: Drug: ETH-155008
  Interventions: Drug: ETH-155008

INTERVENTIONS:
Drug: ETH-155008 — ETH-155008 is an orally bioavailable, potent Pim-3 and CDK4/6 dual kinase inhibitor.
  Dosage form: 10mg, 20 mg and 40 mg, tablets. ETH-155008 tablets should be taken while fasting, either 1 hour before or 2 hours after a meal.
  Other Names: Study drug

SUMMARY:
This Trial is an open-label, multicenter trial to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of ETH-155008 in subjects with AML and NHL who previously received standard treatment or are ineligible for standard treatment options.

DETAILED DESCRIPTION:
The primary objectives of this study are to evaluate the safety of ETH-155008 and to determine the recommended Phase 2 dose (RP2D) regimen or the maximum tolerated dose (MTD). Secondary objectives and endpoints will evaluate the pharmacokinetics(PK) and pharmacodynamics(PD) of ETH-155008 and preliminary clinical anti-tumor activity of ETH-155008 in subjects with R/R acute myeloid leukemia (AML) and Non-Hodgkin's lymphoma (NHL).

This Trial is an open-label, multicenter trial to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of ETH-155008 in subjects with R/R AML and NHL who previously received standard treatment or are ineligible for standard treatment options. The study will be conducted in 2 parts: dose escalation (Part 1) and cohort expansion (Part 2). In the dose escalation, ETH-155008 will be administrated orally, once daily (QD) for 28 days at 5 dose levels ranging from 20 mg to 100 mg in 28-day cycles. Dose-limiting toxicity (DLT) will be assessed during the first treatment cycle and the maximum tolerated dose (MTD) will be identified. Additional subjects will be treated in the dose expansion at the commended phase 2 dose (RP2D).

During the study, safety will be monitored by the data review committee (DRC) at each dose escalation step and at regular intervals during cohort expansion. Continuous reassessment for DLTs will help minimize the potential risks associated with the study drug. Cumulative data from subsequent treatment cycles will also be monitored for late-onset toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age and < 80 years old.
2. Must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the trial and are willing to participate in the trial prior to any other trial-related assessments or procedures, and can communicated with investigators and are willing to comply with the protocol.
3. Has histologically or cytologically confirmed relapsed and/or refractory acute myelocytic leukemia(AML) or non-Hodgkin's lymphoma(NHL) with no available standard therapy or is not a candidate for available standard therapy, and for whom, in the opinion of the investigator, experimental therapy with ETH-155008 may be beneficial. In addition, the following disease-specific criteria outlined below must be met.

   1. For all indolent NHL (Follicular Lymphoma[FL], Marginal Zone Lymphoma[MZL] and Waldenström Macroglobulinemia[WM]), previously treated with at least 2 prior lines of systemic therapy with at least 1 line being an anti-cluster of differentiation antigen 20(anti-CD20) antibody-containing combination regimen. For chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), prior treatment with at least 2 lines of systemic therapy, including Bruton's tyrosine kinase(BTK) inhibitors or B-cell lymphoma-2(BCL-2) inhibitors, is required.
   2. For mantle cell lymphoma(MCL), prior treatment with at least 2 lines of systemic therapy (including a combination regimen of anti-CD20 antibodies and BTK inhibitors) and no other approved therapy considered more appropriate by the investigators.
   3. For aggressive B-NHL (diffuse large B cell lymphoma[DLBCL], highly malignant B-cell lymphoma[HGBCL], and primary mediastinal large B-cell lymphoma[PMBCL]), patients who can tolerate intensive therapy or autologous hematopoietic stem cell transplantation are required to have received standard second-line therapy in the past but have failed or relapsed. If patients cannot tolerate intensive therapy or autologous hematopoietic stem cell transplantation, they must have received standard first-line therapy in the past, but therapy failed or relapsed.
   4. For T-NHL, it is required to have been adequately treated with a systemic standard dose of drugs in the past without remission or recurrence.
   5. For AML, relapsed/refractory AML diagnosed according to the World Health Organization (WHO) classification in 2016, for which no standard treatment is available or for which standard treatment is not tolerated; According to Chinese Guidelines for the Diagnosis and Treatment of Relapsed and Refractory acute myeloid Leukemia (2021 Edition), the definition of relapsed and refractory is as follows:

   <!-- -->

   1. Recurrent AML: recurrence of leukemia cells in peripheral blood or original cells in bone marrow ≥ 5% after CR (except for other reasons such as bone marrow regeneration after consolidation chemotherapy) or extramedullary leukemia cell infiltration.
   2. Refractory AML: initial patients who failed to respond to 2 courses of treatment with standard protocols; Patients with CR relapse within 12 months after consolidation and intensive treatment; Patients who relapse after 12 months but fail to respond to conventional chemotherapy; Patients with two or more relapses; Extramedullary leukemia persists.
4. For NHL, measurable lesions that meet the efficacy evaluation criteria for Lugano lymphoma (Cheson 2014) are required(at least one intranodular lesion longest diameter (LDi)﹥1.5 cm, or at least 1 extranodal lesion LDi﹥1 cm). For WM patients, immunoglobulin M(IgM) should be greater than 5g/L. For chronic lymphocytic leukemia(CLL) patients, monoclonal B lymphocytes greater than 5×109/L are required. For patients with AML, bone marrow primordial cells at baseline are required to be at least 5%.
5. Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1 (dose escalation cohorts) or ≤2 (dose expansion cohorts).
6. For NHL, hematology laboratory parameters must be within the following ranges. Values must be without transfusions or growth factors for at least 7 days prior to the first dose of study drug ,

   1. Hemoglobin (HB) ≥80g/L; In case of bone marrow invasion, hemoglobin ≥60g/L is required (red blood cell infusion is allowed prior to initial administration).
   2. Platelet (PLT) count ≥75×10^9/L; In case of bone marrow invasion, platelet count ≥50×10^9/L (50,000/μL) is required.
   3. Absolute count of neutrophil granulocyte (ANC) ≥1.0×10^9/L; Absolute neutrophil count ≥0.75×10^9/L (750/μL) is required if bone marrow invasion is present.
7. For AML, there is no upper limit on white blood cell count (WBC) at screening, but it is required before the first administration of the investigational drug WBC﹤25×10^9/L. Note: Subjects with excess primitive cells may be treated with hydroxyurea until 2 days prior to initial administration of the study drug to reduce WBC.
8. Blood biochemical test results must be within the following range:

   1. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5×upper limit of normal (ULN). If the subject has primary liver invasion, ALT, AST ≤5×ULN is required.
   2. Total bilirubin(TBIL) ≤1.5×ULN. If the subject has primary liver invasion, TBIL ≤3×ULN is required.
   3. Creatinine clearance rate(CCr)≥45 ml/min (Cockcroft-Gault formula).
   4. Prothrombin time(PT) and activated partial thromboplastin time(aPTT) ≤1.5×ULN.
9. Life expectancy of at least 3 months.
10. A woman of childbearing potential must have a negative serum beta-human chorionic gonadotropin (beta-hCG) at screening and prior to the first dose of study drug.
11. Women must be: a. Not of childbearing potential b. Of childbearing potential and - Practicing a highly effective, preferably user-independent method of contraception (failure rate of <1% per year when used consistently and correctly) and agrees to remain on a highly effective method while receiving study drug and until 90 days after last dose.
12. In addition to the user-independent, highly effective method of contraception, a male or female condom is required. Male condoms and female condoms should not be used together (due to risk of failure with friction).
13. A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control, e.g., either condom with or partner with occlusive cap (diaphragm or cervical/vault caps).
14. Men or women must agree not to donate sperm or eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 3 months after the last study drug administration.
15. Must be willing and able to adhere to the requirements and restrictions specified in the ICF and this protocol.

Exclusion Criteria:

1. Acute promyelocytic leukemia, acute mixed phenotypic leukemia, acute myeloid leukemia with Philadelphia chromosome (Ph chromosome) positive.
2. AML with myeloid sarcoma.
3. The central nervous system (CNS) is known to be involved.
4. Previous solid organ transplantation.
5. Previously received allogeneic hematopoietic stem cell transplantation.
6. The patient received autologous hematopoietic stem cell transplantation (HSCT) within 3 months prior to initial administration of ETH-155008.
7. Have an active autoimmune disease within the past 2 years that requires treatment with systemic immunosuppressive drugs (i.e., long-term corticosteroids, methotrexate, or tacrolimus).
8. Toxicities from previous anti-cancer therapies have not resolved to baseline levels or to Grade 1 or less except for alopecia and peripheral neuropathy.
9. Has known past or current malignancy other than inclusion diagnosis, except for:

   1. Cervical carcinoma of Stage ⅠB or less.
   2. Non-invasive basal cell or squamous cell skin carcinomas.
   3. Non-invasive, superficial bladder cancer.
   4. Prostate cancer with a current prostate-specific antigen(PSA) level < 0.1 ng/mL.
   5. malignancy which in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 1 year before the first dose of study drug.
   6. Any curable cancer with a complete response(CR) of > 2 years duration.
10. Prior treatment with a cyclin dependent kinase 4 and 6(CDK4/6) or Pim inhibitor.
11. Known allergies, hypersensitivity, or intolerance to ETH-155008 or its excipients.
12. Prior chemotherapy or targeted therapy within 2 weeks(Or five half-lives, which is the longer) prior to first dosing treatment, or treatment with an investigational anticancer agent or radiotherapy (including investigational vaccines) within 4 weeks before the first administration of ETH-155008. For investigational agents where half-life is known, there should be a treatment-free window of at least 2 weeks or 5 half-lives.
13. Prior chimeric antigen receptor T-Cell(CAR-T) immunotherapy within 12 weeks before the first administration of ETH-155008.
14. Corticosteroids >10 mg daily prednisone equivalents:

    a. A short course (ie, >10 mg daily prednisone equivalents for less than 7 days) of corticosteroids is permitted. Inhaled or topical steroids, and adrenal replacement doses ≤10 mg daily prednisone equivalents, are permitted in the absence of active autoimmune disease.
15. History of clinically significant cardiovascular disease within the 6 months prior to the first dose of study drug including, but not limited to:

    1. Corrected QT interval (QT interval corrected using Fridericia formula [QTcF]) female﹥470ms, male﹥450ms.
    2. Myocardial infarction
    3. Severe or unstable angina
    4. Clinically significant cardiac arrhythmias
    5. Uncontrolled (persistent) hypertension: systolic blood pressure >159 mmHg; diastolic blood pressure >99 mmHg
    6. Stroke or transient ischemic attack
    7. Venous thromboembolic events (i.e., pulmonary embolism) within 1 month prior to the first dose of study drug
    8. Congestive heart failure (New York Heart Association class III-IV)
    9. Pericarditis or clinically significant pericardial effusion
    10. Myocarditis
    11. Endocarditis
16. Clinically significant pulmonary compromise, particularly the need for supplemental oxygen to maintain adequate oxygenation.
17. Unable to swallow capsules or tablets or malabsorption syndrome, disease significantly affecting GI function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction. If any of these conditions exist, the site should discuss with the sponsor to determine subject eligibility.
18. Evidence of active viral, bacterial, or uncontrolled systemic fungal infection requiring parenteral treatment within 2 weeks before the first dose of study drug.
19. Active or chronic hepatitis B or hepatitis C infection.

    1. Hepatitis B infection is defined by a positive test for hepatitis B surface antigen (HBsAg)
    2. Or HBsAg negative and positive for anti-hepatitis B core antigen (HBc) with hepatitis B virus(HBV) DNA﹥ULN
    3. Hepatitis C infection is defined by a positive hepatitis C virus (HCV) ribonucleic acid (RNA).
20. Tested HIV positive at screening.
21. Syphilitic antibody positive.
22. Trauma or major surgery (e.g., requiring general anesthesia) within 28 days prior to the first dose of study drug. Note: Subjects with planned surgical procedures to be conducted under local anesthesia may participate.
23. Any serious underlying medical or psychiatric condition (e.g., alcohol or drug abuse), dementia or altered mental status; or any issue that would impair the ability of the subject to receive or tolerate the planned treatment at the investigational site, to understand informed consent, or that in the opinion of the investigator would contraindicate the participation in the study or confound the protocol-specified assessments or results of the study.
24. Requires a prohibited medication that cannot be discontinued or substituted, or temporally interrupted during the study.
25. A drug used as a substrate for cytochrome P450 3A4(CYP3A4) within 1 week (or 5 half-lives, whichever was longer) prior to initial treatment.
26. Overactive CYP3A4 or P-glycoprotein inducers or inhibitors were used within 1 week (or 5 half-lives, if older) prior to initial treatment.
27. A woman who is pregnant or breastfeeding.
28. Other patients judged by the investigator to be unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | At the end of Cycle 1 (each cycle is 28 days)
  Determine the safety of ETH-155008 in subjects with R/R AML and NHL
Dose Limiting Toxicity (DLTs) | At the end of Cycle 1 (each cycle is 28 days)
  Incidence of DLTs in the first treatment cycle of ETH-155008
The RP2D(s) or the MTD of ETH-155008 in subjects with R/R AML and NHL | At the end of Cycle 1 (each cycle is 28 days)
  The RP2D is the maximum tolerated dose (MTD) or less.

SECONDARY OUTCOMES:
PK parameter of ETH-155008: Cmax | At the end of Cycle 1 (each cycle is 28 days)
  Maximum Concentration (Cmax) of ETH-155008
PK parameter of ETH-155008: Tmax | At the end of Cycle 1 (each cycle is 28 days)
  Time of First Occurrence of Cmax for ETH-155008
PK parameter of ETH-155008: AUC | At the end of Cycle 1 (each cycle is 28 days)
  area under the curve (AUC)
Disease evaluation of efficacy of ETH-155008: ORR | 12 months post first dosing
  objective response rate(ORR)
Disease evaluation of efficacy of ETH-155008: CR | 12 months post first dosing
  complete response(CR)
Disease evaluation of efficacy of ETH-155008: PR | 12 months post first dosing
  partial response(PR)
Disease evaluation of efficacy of ETH-155008: DCR | 12 months post first dosing
  disease control rate(DCR)
Disease evaluation of efficacy of ETH-155008: TTR | 12 months post first dosing
  time to response(TTR)
Disease evaluation of efficacy of ETH-155008: DOR | 12 months post first dosing
  duration of response(DOR)
Assess the PD of ETH-155008: Inhibition of Pim kinase | 2 months post first dosing
  Inhibition of Pim kinases
Assess the PD of ETH-155008: Inhibition of CDK4/6 kinase | 2 months post first dosing
  Inhibition of cyclin-dependent kinase 4 and 6(CDK4/6)
Assess the PD of ETH-155008: Inhibition of FLT3 kinase | 2 months post first dosing
  Inhibition of Feline McDonough sarcoma-like tyrosine kinase 3(FLT3)

CONTACTS AND LOCATIONS:
Overall Officials: James Zhang, Study Director — Shengke Pharmaceuticals (Jiangsu) Limited, China
Locations (2):
- China (2):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hematology Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No